CLINICAL TRIAL: NCT02268318
Title: A RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, PARALLEL STUDY TO EVALUATE THE EFFECT OF A 12-WEEK CONSUMPTION PERIOD OF SINGLE DOSE A DAY OF A PLANT STEROL-ENRICHED FERMENTED DAIRY PRODUCT ON BLOOD LIPOPROTEIN PROFILE IN JAPANESE ADULTS WITH HIGH LDL-C
Brief Title: "A Clinical Study for Evaluating the Effect of a Plant Sterol-enriched Fermented Dairy Product on Blood Lipoprotein Profile in Japanese Adults"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Japan (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: NU359
Record Dates: First submitted 2014-10-16; First posted 2014-10-20 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Subjects With High LDL-Cholesterol
Keywords: Japanese Subjects, High LDL-C, fermented-dairy products, phytosterols
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1-Fermented Dairy Product with Phytosterols (test) (Experimental): one arm active = 1 bottle of dairy product/day with 1,6g of phytosterols
  Interventions: Other: 1-Fermented Dairy Product with Phytosterols (test)
- 2-Fermented dairy Product with No Phytosterols (control) (Placebo Comparator): one arm control product= 1 bottle of dairy product/day with no Phytosterols
  Interventions: Other: 2-Fermented dairy Product with No Phytosterols (control)

INTERVENTIONS:
Other: 1-Fermented Dairy Product with Phytosterols (test) — 1- 1 bottle of test product/day
  Arms: 1-Fermented Dairy Product with Phytosterols (test)
Other: 2-Fermented dairy Product with No Phytosterols (control) — 2-1 bottle of control product/day
  Arms: 2-Fermented dairy Product with No Phytosterols (control)

SUMMARY:
INVESTIGATE THE EFFECT OF A 12-WEEK CONSUMPTION PERIOD OF SINGLE DOSE A DAY OF A PLANT STEROLS-ENRICHED FERMENTED DAIRY PRODUCT ON BLOOD LIPOPROTEIN PROFILE IN JAPANESE ADULTS WITH HIGH LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* An individual must fulfil all of the following criteria in order to be eligible for trial enrolment

To be checked at the inclusion visit (V1):

* II 01: Male/female subject, aged from 20 to 75 years (bounds included).
* II 02: Subject with body mass index (BMI) between 18.5 kg/m2 (bound included) and 30 kg/m2 (bound excluded).
* II 03: Subject with LDL-cholesterol blood level between 120 mg/dL (3.1 mmol/L) and 160 mg/dL (4.14 mmol/L) (bounds included).
* II 04: Subject with triglycerides under 200 mg/dL (2.3 mmol/L).
* II 05: Non hypertensive subject defined with Systolic Blood Pressure (SBP) <140 mmHg and Diastolic Blood Pressure (DBP) <90 mmHg OR subject with treated and controlled hypertension defined with SBP <140 mmHg and DBP <90 mmHg since at least 1 month.
* II 06: Subject who already received the dietary recommendations advisable for hyper or borderline hyper-LDL cholesterolemic subjects (according to Japan Atherosclerosis Society guidelines).
* II 07: Subject agreeing not to consume any supplements/ food products enriched with plant sterols and plant stanols in any form and soy milk product during the study period.
* II 08: Female subject must be postmenopausal for at least 12 months prior to trial entry or surgically sterile (i.e. hysterectomy, bilateral oophorectomy or bilateral tubal ligation) OR if of child bearing potential, female subject must be using or complying with one of the following medically approved methods of contraception such as, but not exclusively:
* Oral birth control pills (at least 1 full monthly cycle prior to study product administration);
* Intra-uterine device (IUD);
* Double barrier methods (such as condoms and spermicide);
* Abstinence, when in the opinion of the investigator, their occupation or life style gives efficient evidence that abstinence will be maintained throughout the study and for one month thereafter.
* II 09: Subject covered by social security or covered by similar system.
* II 10: Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective; and being able to personally sign a written informed consent.
* II 11: Subject having given written (dated and signed) inform consent to take part in the study.
* II 12: Asian subjects originating from Japan.
* II 13: Subject who is able to communicate well with the investigator and to comply with the requirements of the entire study.
* II 14: Subject having a fridge at home for study products storage with sufficient capacity.

To be checked at the randomization visit (V2):

* RI 01: Subject with LDL-cholesterol blood level between 120 mg/dL (3.1 mmol/L) and 160 mg/dL (4.14 mmol/L) (bounds included).
* RI 02: Subject with triglycerides under 200 mg/dL (2.3 mmol/L).
* RI 03: Subject having compliance to the product during the run-in period 80%.
* RI 04: Subject having followed the dietary recommendations advisable for hypercholesterolaemic patients.

Exclusion Criteria:

* An individual fulfilling any of the following criteria is to be excluded from trial enrolment

To be checked at the inclusion visit (V1):

* IE 01: Subject under hypocholesterolaemic treatment.
* IE 02: Subjects having stopped taking their hypocholesterolemic drugs or products (statins, ezetimibe, sequesterants, niacin, nicotinates, probucol, omega-3 fatty acids (EPA-DHA, ALA…), and fibrates) less than 3 months ago.
* IE 03: Subject with known allergy or hypersensitivity to plant sterols and to any component of the study product (milk protein for example).
* IE 04: Subjects having sitosterolemia.
* IE 05: Subject having experienced any cardiovascular event (cardiac infarction, angina attack, surgical or endoscopic coronary angioplasty, stroke, arterial disease, etc.).
* IE 06: Subject suffering from any serious or chronic liver, renal, cardiovascular, respiratory, endocrine or metabolic disorders.
* IE 07: Subject with gastro-intestinal disorders (such as diarrhoea, constipation, irritable bowel syndrome) or using laxatives.
* IE 08: Subject with diabetes Type I and Type II or Fasting Blood Sugar test (FBS) > 125 mg/dL (7.0 mmol/L) at screening visit.
* IE 09: Subject who had any surgery or intervention requiring a general anesthesia in the preceding 4 weeks, or who plans to have one during the course of the study.
* IE 10: Subject receiving (currently or in the 4 last weeks) systemic treatment or topical treatment likely to interfere with evaluation of the study parameters.
* IE 11: Subject involved in any other clinical study within the preceding month or in the exclusion period after another clinical study.
* IE 12: Subject having blood sample of 200 mL or more taken (e.g., donated blood) within 1 month, or 400 mL or more within 3 months before the start of the present study.
* IE 13: Subject with heavy alcohol intake (> 60 g/day).
* IE 14: Subject taking any treatment for anorexia, weight loss, or any form of treatment likely to interfere with metabolism or dietary habits (e.g. hypolipemic, hypoglycaemic treatments).
* IE 15: For female subject: pregnant woman or woman planning to become pregnant during the study; breast-feeding woman.
* IE 16: For female subject: subject likely to change her contraceptive method or hormone replacement therapy during the study.
* IE 17: Subject in a situation, which in the investigator's opinion could interfere with optimal participation in the present study (e.g. non-dairy-products consumer) or could constitute a special risk for the subject.
* IE 18: Subject who is susceptible to not comply with dietary qualitative restriction during the study period.
* IE 19: Vulnerable subjects defined as individuals whose willingness to volunteer in the clinical trial may be unduly influenced by the expectation, whether justified or not, of benefits associated with participation, or of a retaliatory response from senior members of a hierarchy in case of refusal to participate. Examples are members of a group with a hierarchical structure, such as medical, pharmacy, dental and nursing students, subordinate hospital and laboratory personnel, employees of the pharmaceutical industry, members of the armed forces, and persons kept in detention.
* IE 20: Subjects with known lactose intolerance or known allergy to plant sterols.
* IE 21: Subjects being a heavy soybean milk consumer.
* IE 22: Subject expected to be living in the same home as a current participating subject and to concomitantly receive some study products.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Evolution of LDL-cholesterol concentration after 6 weeks of product consumption, expressed as a relative change from baseline. | baseline and 6 weeks

SECONDARY OUTCOMES:
- Evolution of LDL-cholesterol concentration after 6 weeks of product consumption, expressed as a raw change from baseline. - Evolution of LDL-cholesterol concentration after 3 and 12 weeks of product consumption, expressed as a relative and raw changes | baseline, 3 / 6 / 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christine MRINI, MD, PHD, Study Director — Danone Research Life Sciences
Locations (1):
- Yaesu Sakura-dori Clinic, Tokyo, Japan